CLINICAL TRIAL: NCT02815579
Title: Agricultural Intervention for Food Security and HIV Health Outcomes in Kenya
Acronym: Shamba R01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kenya Medical Research Institute (Other); University of South Carolina (Other); University of Connecticut (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P0503135; R01MH107330-01 (NIH)
Record Dates: First submitted 2016-05-11; First posted 2016-06-28 (Estimated); Results first posted 2024-01-18 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: HIV
Keywords: HIV; Food insecurity; Microcredit loan; Agriculture; Livelihoods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Shamba Maisha Intervention includes: a) a loan (~$175) from a well-established Kenyan bank for purchasing agricultural implements and commodities; b) agricultural implements to be purchased with the loan including the KickStart treadle pump, seeds, fertilizers and pesticides; and c) education in financial management and sustainable farming practices occurring in the setting of patient support groups.
  Interventions: Other: Shamba Maisha Intervention
- Control (No Intervention): Participants in the control arm will receive the standard of care.

INTERVENTIONS:
Other: Shamba Maisha Intervention — A) A loan (~$175) B) Agricultural implements to be purchased with the loan C) Education in financial management and sustainable farming practices
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether this multisectoral agricultural and microcredit loan intervention improves food security, prevent antiretroviral treatment failure, and reduce co-morbidities among people living with HIV/AIDS.

DETAILED DESCRIPTION:
Despite major advances in care and treatment for those living with HIV, morbidity and mortality among people living with HIV/AIDS (PLHIV) remains unacceptably high in sub-Saharan Africa (SSA), largely due to the parallel challenges of poverty and food insecurity.[1] In the Nyanza Region of Kenya, 15.1% of the adult population is infected by HIV,[2] and over 50% of the rural population is food insecure, primarily due to unpredictable rainfall and limited irrigation.[3,4] The investigators have previously shown that food insecurity delays antiretroviral therapy (ART) initiation, reduces ART adherence, contributes to worse immunologic and virologic outcomes, and increases morbidity and mortality among PLHIV.[5-16] There has been increasing international recognition that improved food security and reduced poverty are essential components for a successful global response to the HIV epidemic.[17-21] Yet, to date few studies have systematically evaluated the impacts of sustainable food security interventions on health, economic, and behavioral outcomes among PLHIV. Agricultural interventions, which have potential to raise income and bolster food security, are an important but understudied route through which to sustainably improve nutritional and HIV outcomes in SSA, including Kenya where agriculture accounts for > 75% of the total workforce, and 51% of the gross domestic product.[22]

Building on the investigators successful completion of the pilot intervention trial in Kenya and the investigators collective experience studying structural barriers to HIV care in SSA, the investigators plan to test the hypothesis that a multisectoral agricultural and microcredit loan intervention will improve food security, prevent ART treatment failure, and reduce co-morbidities among PLHIV. The investigators' intervention was co-developed with KickStart, a prominent non-governmental organization (NGO) based in SSA that has introduced a human-powered pump, enabling farmers to grow high yield crops year-round. This technology has reduced food insecurity and poverty for 800,000 users in 22 countries in the subcontinent since 1991.[23] The investigators' intervention includes: a) a loan (~$175) from a well-established Kenyan bank for purchasing agricultural implements and commodities; b) agricultural implements to be purchased with the loan including the KickStart treadle pump, seeds, fertilizers and pesticides; and c) education in financial management and sustainable farming practices occurring in the setting of patient support groups. This study is a cluster randomized controlled trial (RCT) of this intervention with the following specific aims:

Aim 1: To determine the impact of a multisectoral agricultural intervention among HIV-infected farmers on ART on HIV clinical outcomes. The investigators hypothesize that the intervention will lead to improved viral load suppression (primary outcome) and changes in CD4 cell count, physical health status, WHO stage III/IV disease, and hospitalizations (secondary outcomes) in the intervention arm compared to the control arm.

Aim 2: To understand the pathways through which the multisectoral intervention may improve HIV health outcomes. Using the investigator's theoretical model,[1,24] the investigators hypothesize that the intervention will improve food security and household wealth, which in turn will contribute to improved outcomes through nutritional (improved nutritional status measured with Body Mass Index), behavioral (improved ART adherence, and retention in care), and mental health (improved mental health/less depression, improved empowerment) pathways (secondary outcomes).

Aim 3: To determine the cost-effectiveness of the intervention and obtain the information necessary to inform scale-up in Kenya and similar settings in SSA. The investigators will quantify the cost per disability-adjusted life year averted, and identify lessons to inform successful scale-up.

To accomplish Aims 1 & 2, the investigators will randomize 8 matched pairs of health facilities in the Nyanza Region in a 1:1 ratio to the intervention and control arms, and enroll 44 participants per facility (total n=704). All participants will be followed for 2 years. Impacts of the investigator's intervention on primary health outcomes and mediators will be investigated to provide definitive data of direct and indirect intervention effects. To accomplish Aim 3, the investigators will: a) conduct a cost-effectiveness analysis; b) identify the characteristics of individuals most likely to benefit from the intervention (e.g., gender, educational attainment, family size, wealth, risk tolerance, and entrepreneurial ability); and c) perform a mixed-methods process evaluation with study participants, staff, and various stakeholders to determine what worked and did not work to guide future scale-up efforts of the intervention.

The investigator's ultimate goal is to develop and test an intervention to reverse the cycle of food insecurity and HIV/AIDS morbidity and mortality in SSA.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected adults
* Currently receiving ART
* Belong to a patient support group or demonstrate willingness to join a support group
* Agree to save the down payment (~$10) required for the microcredit loan
* Have evidence of moderate to severe food insecurity based on the Household Food Insecurity Access Scale (HFIAS), and/or malnutrition (BMI<18.5) based on FACES medical records during the year preceding recruitment
* Have access to farming land and available surface water in the form of lakes, rivers, ponds and shallow wells

Exclusion Criteria:

* People who do not speak Dholuo, Swahili, or English
* Inadequate cognitive and/or hearing capacity to complete planned study procedures, at the discretion of the research assistant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 746 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheri D Weiser, MD, MPH, Principal Investigator — Departments of Medicine, UCSF; Craig R Cohen, MD, MPH, Principal Investigator — Department of Obstetrics, Gynecology & Reproductive Sciences, UCSF
Locations (16):
- Kenya (16):
  - Kitare, Suba, Homa Bay County
  - Sindo, Suba, Homa Bay County
  - Muhuru Bay, Nyatike, Migori County
  - Sori Lakeside, Nyatike, Migori County
  - Minyenya, Rongo, Migori County
  - Ngode, Rongo, Migori County
  - Oyani, Rongo, Migori County
  - Nyamasare, Uriri, Migori County
  - Hongo Ogosa, Kisumu
  - Kisumu District Hospital, Kisumu
  - Lumumba, Kisumu
  - Nyangande, Kisumu
  - Pandiperi, Kisumu
  - Railways, Kisumu
  - Osingo, Migori
  - Suna Ragana, Migori

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiser SD, Young SL, Cohen CR, Kushel MB, Tsai AC, Tien PC, Hatcher AM, Frongillo EA, Bangsberg DR. Conceptual framework for understanding the bidirectional links between food insecurity and HIV/AIDS. Am J Clin Nutr. 2011 Dec;94(6):1729S-1739S. doi: 10.3945/ajcn.111.012070. Epub 2011 Nov 16. PMID 22089434
- [Background] National AIDS and STI Control Programme, Ministry of Health, Kenya. September 2013. Kenya AIDS Indicator Survey 2012: Preliminary Report. Nairobi, Kenya
- [Background] Place F, Adato M, Hebinck P. Understanding rural poverty and investment in agriculture: an assessment of integrated quantitative and qualitative research in western Kenya. World Dev. 2007;35(2):312-325.
- [Background] Stoorvogel J, Smaling E. Assessment of soil nutrient depletion in sub-Saharan Africa: 1983-2000. Report No. 28, Vols. I-IV. Wageningin, Netherlands: Winand Staring Center; 1990.
- [Background] McMahon JH, Wanke CA, Elliott JH, Skinner S, Tang AM. Repeated assessments of food security predict CD4 change in the setting of antiretroviral therapy. J Acquir Immune Defic Syndr. 2011 Sep 1;58(1):60-3. doi: 10.1097/QAI.0b013e318227f8dd. PMID 21694604
- [Background] Wang EA, McGinnis KA, Fiellin DA, Goulet JL, Bryant K, Gibert CL, Leaf DA, Mattocks K, Sullivan LE, Vogenthaler N, Justice AC; VACS Project Team. Food insecurity is associated with poor virologic response among HIV-infected patients receiving antiretroviral medications. J Gen Intern Med. 2011 Sep;26(9):1012-8. doi: 10.1007/s11606-011-1723-8. Epub 2011 May 15. PMID 21573882
- [Background] Weiser SD, Palar K, Frongillo EA, Tsai AC, Kumbakumba E, Depee S, Hunt PW, Ragland K, Martin J, Bangsberg DR. Longitudinal assessment of associations between food insecurity, antiretroviral adherence and HIV treatment outcomes in rural Uganda. AIDS. 2014 Jan 2;28(1):115-20. doi: 10.1097/01.aids.0000433238.93986.35. PMID 23939234
- [Background] Nagata JM, Magerenge RO, Young SL, Oguta JO, Weiser SD, Cohen CR. Social determinants, lived experiences, and consequences of household food insecurity among persons living with HIV/AIDS on the shore of Lake Victoria, Kenya. AIDS Care. 2012;24(6):728-36. doi: 10.1080/09540121.2011.630358. Epub 2011 Dec 7. PMID 22150119
- [Background] Weiser SD, Tsai AC, Gupta R, Frongillo EA, Kawuma A, Senkungu J, Hunt PW, Emenyonu NI, Mattson JE, Martin JN, Bangsberg DR. Food insecurity is associated with morbidity and patterns of healthcare utilization among HIV-infected individuals in a resource-poor setting. AIDS. 2012 Jan 2;26(1):67-75. doi: 10.1097/QAD.0b013e32834cad37. PMID 21904186
- [Background] Young S, Wheeler AC, McCoy SI, Weiser SD. A review of the role of food insecurity in adherence to care and treatment among adult and pediatric populations living with HIV and AIDS. AIDS Behav. 2014 Oct;18 Suppl 5(0 5):S505-15. doi: 10.1007/s10461-013-0547-4. PMID 23842717
- [Background] Weiser SD, Gupta R, Tsai AC, Frongillo EA, Grede N, Kumbakumba E, Kawuma A, Hunt PW, Martin JN, Bangsberg DR. Changes in food insecurity, nutritional status, and physical health status after antiretroviral therapy initiation in rural Uganda. J Acquir Immune Defic Syndr. 2012 Oct 1;61(2):179-86. doi: 10.1097/QAI.0b013e318261f064. PMID 22692093
- [Background] Weiser S, Fernandes K, Anema A, et al. Food insecurity as a barrier to antiretroviral therapy (ART) adherence among HIV-infected individuals in British Columbia. 5th IAS Conference on HIV Pathogenesis, Treatment and Prevention. Cape Town, South Africa2009.
- [Background] Weiser SD, Fernandes KA, Brandson EK, Lima VD, Anema A, Bangsberg DR, Montaner JS, Hogg RS. The association between food insecurity and mortality among HIV-infected individuals on HAART. J Acquir Immune Defic Syndr. 2009 Nov 1;52(3):342-9. doi: 10.1097/QAI.0b013e3181b627c2. PMID 19675463
- [Background] Musumari PM, Feldman MD, Techasrivichien T, Wouters E, Ono-Kihara M, Kihara M. "If I have nothing to eat, I get angry and push the pills bottle away from me": A qualitative study of patient determinants of adherence to antiretroviral therapy in the Democratic Republic of Congo. AIDS Care. 2013;25(10):1271-7. doi: 10.1080/09540121.2013.764391. Epub 2013 Feb 6. PMID 23383757
- [Background] Musumari PM, Wouters E, Kayembe PK, Kiumbu Nzita M, Mbikayi SM, Suguimoto SP, Techasrivichien T, Lukhele BW, El-Saaidi C, Piot P, Ono-Kihara M, Kihara M. Food insecurity is associated with increased risk of non-adherence to antiretroviral therapy among HIV-infected adults in the Democratic Republic of Congo: a cross-sectional study. PLoS One. 2014 Jan 15;9(1):e85327. doi: 10.1371/journal.pone.0085327. eCollection 2014. PMID 24454841
- [Background] Sasaki Y, Kakimoto K, Dube C, Sikazwe I, Moyo C, Syakantu G, Komada K, Miyano S, Ishikawa N, Kita K, Kai I. Adherence to antiretroviral therapy (ART) during the early months of treatment in rural Zambia: influence of demographic characteristics and social surroundings of patients. Ann Clin Microbiol Antimicrob. 2012 Dec 28;11:34. doi: 10.1186/1476-0711-11-34. PMID 23270312
- [Background] Byron E, Gillespie S, Nangami M. Integrating nutrition security with treatment of people living with HIV: lessons from Kenya. Food Nutr Bull. 2008 Jun;29(2):87-97. doi: 10.1177/156482650802900202. PMID 18693472
- [Background] The World Bank. HIV/AIDS, Nutrition, and Food Security: What we can do. Washington DC2007.
- [Background] UNAIDS. Report on the global AIDS epidemic. Geneva: Joint United Nations Programme on HIV/AIDS;2008.
- [Background] World Health Organization. HIV, food security, and nutrition: World Food Program, UNAIDS;2008.
- [Background] Mamlin J, Kimaiyo S, Lewis S, Tadayo H, Jerop FK, Gichunge C, Petersen T, Yih Y, Braitstein P, Einterz R. Integrating nutrition support for food-insecure patients and their dependents into an HIV care and treatment program in Western Kenya. Am J Public Health. 2009 Feb;99(2):215-21. doi: 10.2105/AJPH.2008.137174. Epub 2008 Dec 4. PMID 19059851
- [Background] USAID. Feed the Future Program, country profile for Kenya. http://www.feedthefuture.gov/country/kenya. Accessed August 4, 2014.
- [Background] KickStart. KickStart Impact. http://www.kickstart.org/what-we-do/impact/. Accessed July 11, 2014.
- [Background] Weiser S, Palar K, Hatcher A, S. Y, Frongillo EA, Laraia BA. Food insecurity and health: A Conceptual Framework. In: Ivers L, ed. Food Insecurity and Public Health. Boston, MA: CRC Press; 2014.
- [Derived] Nicastro TM, Mocello AR, Weke E, Bukusi EA, Frongillo EA, Cohen CR, Weiser SD, Kadiyala S, Harris-Fry HA. Effect of a climate-smart intervention on agriculture and nutrition of people with HIV. AIDS. 2025 Sep 1;39(11):1650-1655. doi: 10.1097/QAD.0000000000004234. Epub 2025 May 14. PMID 40372058
- [Derived] Richards AL, Hiepler AJ, Frongillo EA, Khan S, Holding P, Nanga K, Kammerer B, Otieno P, Butler LM. Influence of recurrent assessments during data collection on caregivers and young children for an agricultural livelihood intervention in Kenya: a qualitative study. BMJ Open. 2024 Jun 8;14(6):e077637. doi: 10.1136/bmjopen-2023-077637. PMID 38851226
- [Derived] Sheira LA, Wekesa P, Cohen CR, Weke E, Frongillo EA, Mocello AR, Dworkin SL, Burger RL, Weiser SD, Bukusi EA. Impact of a livelihood intervention on gender roles and relationship power among people with HIV. AIDS. 2024 Jan 1;38(1):95-104. doi: 10.1097/QAD.0000000000003742. Epub 2023 Sep 29. PMID 37788108
- [Derived] Cohen CR, Weke E, Frongillo EA, Sheira LA, Burger R, Mocello AR, Wekesa P, Fisher M, Scow K, Thirumurthy H, Dworkin SL, Shade SB, Butler LM, Bukusi EA, Weiser SD. Effect of a Multisectoral Agricultural Intervention on HIV Health Outcomes Among Adults in Kenya: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2246158. doi: 10.1001/jamanetworkopen.2022.46158. PMID 36508217
- [Derived] Miller JD, Frongillo EA, Weke E, Burger R, Wekesa P, Sheira LA, Mocello AR, Bukusi EA, Otieno P, Cohen CR, Weiser SD, Young SL. Household Water and Food Insecurity Are Positively Associated with Poor Mental and Physical Health among Adults Living with HIV in Western Kenya. J Nutr. 2021 Jun 1;151(6):1656-1664. doi: 10.1093/jn/nxab030. PMID 33709134
- [Derived] McDonough A, Weiser SD, Daniel A, Weke E, Wekesa P, Burger R, Sheira L, Bukusi EA, Cohen CR. "When I Eat Well, I Will Be Healthy, and the Child Will Also Be Healthy": Maternal Nutrition among HIV-Infected Women Enrolled in a Livelihood Intervention in Western Kenya. Curr Dev Nutr. 2020 Mar 13;4(4):nzaa032. doi: 10.1093/cdn/nzaa032. eCollection 2020 Apr. PMID 32270133

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Health Facilities
Groups:
- Intervention: Participants received the Shamba Maisha Intervention that includes: a) a loan (~$175) from a well-established Kenyan bank for purchasing agricultural implements and commodities; b) agricultural implements to be purchased with the microcredit loan including the KickStart treadle pump, seeds, fertilizers and pesticides; and c) education in financial management and sustainable farming practices occurring in the setting of patient support groups.
- Control: Participants in the control arm received the standard of care (HIV care and treatment only). Participants were eligible for the Shamba Maisha intervention at the end of 2 years of follow-up.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 390; 8 Health Facilities | 356; 8 Health Facilities
Started Study Activities | 366; 8 Health Facilities | 354; 8 Health Facilities
Completed | 344; 8 Health Facilities | 333; 8 Health Facilities
Not Completed | 46; 0 Health Facilities | 23; 0 Health Facilities
Not completed — Non-payment of loan down-payment | 16 | 0
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Moved out of study area before receiving any study activities | 9 | 11
Not completed — Lost to Follow-up | 7 | 4
Not completed — Hospitalized before receipt of any study activities | 1 | 0
Not completed — Uncomfortable with MEMS adherence monitoring cap | 1 | 0
Not completed — Death | 5 | 4
Not completed — Imprisoned | 0 | 2
Not completed — Did not meet enrollment criteria | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all enrolled participants who started study activities. Individuals who were enrolled but who were immediately withdrawn from the study before receiving any study activities were not included in the baseline analysis population.
Groups:
- Intervention: Participants received the multisectoral agricultural intervention.
- Control: Participants in the control arm received the standard of care.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 366 | 354 | 720
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (8.9) | 40.4 (9.3) | 40.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 194 | 396
  Male | 164 | 160 | 324
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Kenyan | 366 | 354 | 720
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 366 | 354 | 720
Currently married [Count of Participants; unit: Participants] | 271 | 251 | 522
Number of people in household [Mean (Standard Deviation); unit: people] | 6.5 (2.6) | 6.1 (2.7) | 6.3 (2.7)
Severely food insecure (vs. moderately) [Count of Participants; unit: Participants] — Food security was measured via the Household Food Insecurity Access Scale (HFIAS)
  Participants | 293 | 275 | 568
BMI <18.5 kg/m^2 [Count of Participants; unit: Participants] | 41 | 45 | 86
CD4+ [Mean (Standard Deviation); unit: cells/mm^3] | 603 (276) | 561 (235) | 582 (257)
Viral load <=200 copies/mL [Count of Participants; unit: Participants] | 314 | 291 | 605
Religion [Count of Participants; unit: Participants]
  Catholic | 363 | 353 | 716
  Muslim | 0 | 1 | 1
  Other religion | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Proportion of Viral Load Suppression (<=200 Copies/mL)
Description: The outcome was the change from baseline to the end of follow-up (2 years) in the proportion of participants in viral load suppression (≤200 copies/mL) compared between study groups using difference-in-differences analyses.
Time Frame: Baseline and endline (2 years after enrollment)
Population: 677 participants who completed endline data collection
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 344 | 333
Participants | 327 | 314
Statistical Analysis 1: Comparison: Intervention vs Control; The investigators produced a difference-in-difference estimate between baseline and year 2 using multi-level logistic regression. Units are in log odds; Test type: Superiority; p = 0.86, Mixed Models Analysis; Difference in log odds = -0.08, 95% CI 2-sided [-1.0 to 0.84]

2. Secondary Outcome: Change (i.e., Linear Trend) in Proportion of Absolute CD4 Count <=500 Cells/mm^3
Description: The outcome was the change (i.e., linear trend) from baseline to the end of follow-up (2 years) of the proportion of participants with a CD4 cell count <=500 cells/mm^3, compared between study groups using difference-in-differences analyses.
Time Frame: Baseline and endline (2 years after enrollment)
Population: 677 participants who completed endline data collection
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 344 | 333
Participants | 128 | 129
Statistical Analysis 1: Comparison: Intervention vs Control; The investigators analyzed longitudinal data measured every 6 months to assess trends in the two study arms and produced a difference-in-differences estimate between baseline and year 2 using multi-level logistic regression. Units are in log odds; Test type: Superiority; p = 0.23, Mixed Models Analysis; Difference in log odds = 0.32, 95% CI 2-sided [-0.28 to 0.92]

3. Secondary Outcome: Change (i.e. Linear Trend) in Mean Physical Health Status
Description: The outcome was the change (i.e. linear trend) from baseline to the end of follow-up (2 years) of the mean physical health score compared between study groups using the differences-in-differences analyses. We used the Medical Outcomes Study HIV Health Survey (MOS-HIV), a tool used to assess health-related quality of life that has been validated in resource-limited settings. Scores standardized to a range of 0 to 100. Higher scores mean a better outcome.
Time Frame: Baseline and endline (2 years after enrollment)
Population: 677 participants who completed endline data collection
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 344 | 333
units on a scale | 86.0 [81.6 to 87.3] | 86.2 [80.5 to 87.6]
Statistical Analysis 1: Comparison: Intervention vs Control; The investigators analyzed longitudinal data measured every 6 months to assess trends in the two study arms and produced a difference-in-differences estimate between baseline and year 2; Test type: Superiority; p = 0.26, Mixed Models Analysis; Mean Difference (Net) = 1.39, 95% CI 2-sided [-1.01 to 3.78]

4. Secondary Outcome: Change (i.e., Linear Trend) in the Proportion of Participants With AIDS-Defining Condition
Description: The outcome was the change (i.e., linear trend) from baseline to the end of follow-up (2 years) of the proportion of participants with an AIDS-defining condition, compared between study groups using difference-in-differences analyses. AIDS-defining conditions including HIV-related illnesses included in the Centers for Disease Control and Prevention's (CDC) list of diagnostic criteria for AIDS. AIDS-defining conditions include opportunistic infections and cancers that are life-threatening in a person with HIV.
Time Frame: Baseline and endline (2 years after enrollment)
Population: 677 participants who completed endline data collection
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 344 | 333
Participants | 4 | 2
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.31, Mixed Models Analysis; Difference in log odds = 0.84, 95% CI 2-sided [-0.79 to 2.47]

5. Secondary Outcome: Change (i.e., Linear Trend) in the Proportion of Participants Who Were Hospitalized in the Previous 6 Months
Description: The outcome was the change (i.e. linear trend) from baseline to end of follow-up (2 years) of the proportion of participants hospitalized in the previous 6 months (yes/no), compared between study groups using difference-in-differences analyses.
Time Frame: Baseline and endline (2 years after enrollment)
Population: 677 participants who completed endline data collection
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 344 | 333
Participants | 21 | 18
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.44, Mixed Models Analysis; Difference in log odds = -0.34, 95% CI 2-sided [-1.22 to 0.53]

6. Secondary Outcome: Change (i.e. Linear Trend) in the Mean Score of Food Insecurity Score
Description: The outcome was the change (i.e. linear trend) from baseline to the end of follow-up (2 years) of the mean household food insecurity score, compared between study groups using difference-in-differences analyses.
  using the Household Food Insecurity Access Scale (HFIAS). The HFIAS is a tool to assess household food insecurity (access). The scale scores range from 0 to 27, with higher scores indicating greater food insecurity.
Time Frame: Baseline and endline (2 years after enrollment)
Population: 677 participants who completed endline data collection
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 344 | 333
score on a scale | 14.0 [11.0 to 18.0] | 15.0 [14.0 to 19.0]
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -3.54, 95% CI 2-sided [-4.16 to -2.92]

7. Secondary Outcome: Change (i.e. Linear Trend) in Mean Nutritional Status (Represented by Body Mass Index (BMI))
Description: The outcome was the change (i.e. linear trend) from baseline to the end of follow-up (2 years) of the mean body mass index (BMI) compared between study grouops using the differences-in-differences analyses.
Time Frame: Baseline and endline (2 years after enrollment)
Population: 677 participants who completed endline data collection
Measure: Mean (Inter-Quartile Range); unit: kg/m^2
Arm/Group | Intervention | Control
Number analyzed (Participants) | 344 | 333
kg/m^2 | 22.1 [20.2 to 24.6] | 21.8 [19.0 to 24.5]
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.02, Mixed Models Analysis; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.39 to -0.04]

8. Secondary Outcome: Change (i.e. Linear Trend) in Mean Self-reported Adherence to Antiretroviral Therapy
Description: The outcome was the change (i.e. linear trend) from baseline to the end of follow-up (2 years) of the mean self-reported adherence to antiretroviral therapy compared between study groups using the differences-in-differences analyses.
Time Frame: Baseline and endline (2 years after enrollment)
Population: 677 participants who completed endline data collection
Measure: Mean (Inter-Quartile Range); unit: percentage of doses taken
Arm/Group | Intervention | Control
Number analyzed (Participants) | 344 | 333
percentage of doses taken | 100 [100 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.98, Mixed Models Analysis; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.82 to 0.84]

9. Secondary Outcome: Change (i.e. Linear Trend) in Mean Self-confidence Score
Description: The outcome was the change (i.e. linear tend) from baseline to the end of follow-up (2 years) in the mean self-confidence score, compared between study groups using difference-in-differences analyses. Self-confidence is measured using the three-item Power Within scale, which has a range of 3 to 9 points where lower scores indicate greater self-confidence.
Time Frame: Baseline and endline (2 years after enrollment)
Population: 677 participants who completed endline data collection
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 344 | 333
score on a scale | 4.0 [4.0 to 6.0] | 4.0 [4.0 to 6.0]
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.37, 95% CI 2-sided [-0.59 to -0.15]

10. Secondary Outcome: Change (i.e. Linear Trend) in Proportion of Probable Depression
Description: The outcome was the change (i.e. linear trend) from baseline to the end of follow-up (2 years) in the proportion with probable depression using the Hopkins Symptom Check-list for Depression, compared between study groups using difference-in-differences analyses.
Time Frame: Baseline and endline (2 years after enrollment)
Population: 677 participants who completed endline data collection
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 344 | 333
Participants | 36 | 41
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.001, Mixed Models Analysis; Difference in log odds = -0.83, 95% CI 2-sided [-1.45 to -0.20]

11. Secondary Outcome: Change (i.e. Linear Trend) in the Mean Internalized Stigma Score
Description: The outcome was the change (i.e. linear trend) from baseline to the end of follow-up (2 years) in the mean internalized stigma score compared between study groups using the differences-in-differences analyses. Internalized HIV stigma arises when someone has accepted and endorsed the negative attitudes towards her/himself due to their HIV status. The internalized HIV stigma sub-scale consisted of six items asking respondents to agree with statements related to how they feel about being HIV positive, such as "having HIV makes me feel like I'm a bad person" and "I feel ashamed of having HIV." Response options ranged from 1 "strongly disagree" to 5 "strongly agree." During the analysis phase, the composite scores of each stigma sub-scale were rescaled to a row average of 1-5, with higher scores indicating greater stigma.
Time Frame: Baseline and endline (2 years after enrollment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 344 | 333
units on a scale | 1.40 (0.68) | 1.72 (0.71)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.42, 95% CI 2-sided [-0.52 to -0.31]

ADVERSE EVENTS:
Time Frame: 2 years
Description: The investigators did not assess participants for serious or other adverse events, other than all-cause mortality.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 5/366 | 4/354
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT02815579/Prot_001.pdf
  • Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT02815579/SAP_002.pdf
  • Informed Consent Form (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT02815579/ICF_000.pdf